CLINICAL TRIAL: NCT04013308
Title: Iontophoresis With Potassium Iodide and the Level of Thyroid Hormones in Healthy Subjects
Brief Title: Iontophoresis With Potassium Iodide and Thyroid Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Jolanta Zwolińska, Head of the Laboratory of Physical Factors, University of Rzeszow
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: URzeszow scientific circle
Record Dates: First submitted 2019-07-03; First posted 2019-07-09 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Thyroid Dysfunction
Keywords: Iontophoresis; potassium iodine; thyroid
MeSH Terms: conditions — Thyroid Diseases | interventions — Iontophoresis; Potassium Iodide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 iontophoresis treatments with potassium iodide (Experimental)
  Interventions: Procedure: Iontophoresis with 2% potassium iodide
- 10 iontophoresis treatments with placebo (No Intervention)

INTERVENTIONS:
Procedure: Iontophoresis with 2% potassium iodide — 10 iontophoresis treatments with 2% potassium iodide on the area of thyroid gland; electrodes with tin foil (Amperage:2mA, duration: 30min)
  Arms: 10 iontophoresis treatments with potassium iodide

SUMMARY:
The aim of the study: To assess the influence of iontophoresis treatment with 2% potassium iodide on the level of thyroid hormones (TSH, FT3, FT4) The study group: conducting 10 iontophoresis treatments with Potassium iodide; The control group: conducting 10 placebo treatments with iontophoresis with destilled water; Intervention: 10 iontophoresis treatments with 2% potassium iodide in healthy individuals.

Test the level of thyroid hormones before and after the 10 iontophoresis treatments; The study allows to assess the influence of iodine on the function of thuroid gland.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals with normal thyroid function

Exclusion Criteria:

* individuals with thyroid disorders,
* taking thyroid medication,
* using drugs, alcohol, cigaretttes

Ages: 19 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
the level of thyroid gland hormones (TSH, FT3, FT4) | change in the thyroid hormones level from the baseline to 14 days after the last treatment
  to test thyroid hormones before and after 10 iontophoresis treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Innovative Research in Medical and Natural Sciences' Medical Faculty of University of Rzeszow, Rzeszów, Podkarpackie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zwolinska J, Augustyn B, Baj K, Krukowska J. The effect of galvanization and potassium iodide iontophoresis of the throat and larynx on thyroid parameters: a randomized controlled trial. Sci Rep. 2021 Aug 2;11(1):15590. doi: 10.1038/s41598-021-95145-w. PMID 34341406